CLINICAL TRIAL: NCT05936957
Title: The Ibadan Acute and Chronic Heart Failure Project
Status: Recruiting | Type: Observational
Sponsor: University College Hospital, Ibadan (Other)
Responsible Party: Principal Investigator, O.S Ogah, Dr, University College Hospital, Ibadan
Other Study IDs: IHFP_Protocol_V1.2_2015; 190371 (Other: University of Ibadan)
Record Dates: First submitted 2022-09-02; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure
Keywords: Heart failure, Cardiac Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute heart failure: These are acutely decompensated heart failure
- Chronic heart failure: These are stable heart failure patients being followed up in the outpatient clinic

SUMMARY:
Contemporary studies from South Africa and Nigeria have built on historical reports to demonstrate that the etiology and indeed case profile of acute HF (i.e. more women and younger individuals affected in the prime of their life) is different from high-income countries. As such, HF is now responsible for 7-10% of medical admissions in the region.

These are entirely based on studies on acute HF and few on chronic HF. The nexus between endemic infections such as tuberculosis (TB) and HIV/AIDS and other non-communicable or non-infectious risk factors and HF in Africa is scarcely documented.

This study will assess the long-term outcomes, risk factors, clinical phenotypes, and genomics of HF in Ibadan, Nigeria, estimate catastrophic healthcare cost associated with CHF and how it affects evidence-based care; understand cultural and social conceptions of HF in the city and by extension in Nigeria.

Data from each subject shall be obtained using a uniform and standardized case report forms (CRF). A detailed clinical documentation on cases of HF will be undertaken.

All variables will be summarized using appropriate descriptive statistics. Means and proportions will be estimated with two-tailed 95% confidence intervals. Specified patients' outcomes will also be summarized using proportions. Factors associated wit patient outcomes will be investigated using multivariable logistic regression models. Crude and adjusted Odds Ratio (OR) with 95% confidence intervals (CI) will be estimated.

The primary event outcome of the study will be mortality by cause. Secondary event outcomes will include non-fatal major events (both resulting in and not resulting in admission).

DETAILED DESCRIPTION:
Background and Purpose Heart failure (HF) has emerged a major global public health problem.(1,2) HF affects over 64 million people worldwide. (3) It is a highly symptomatic syndrome that affects 2-3% of the population in high income countries especially in people above the age of 65 years. (4 5) Until recently, little was known about the emerging problem of non-communicable forms of HF supplementing traditional pathways to the syndrome in sub-Saharan Africa due to infections and infestations. Contemporary studies from South Africa (6) and Nigeria (7) have built on historical reports to demonstrate that the aetiology and indeed case profile of acute HF (i.e. more women and younger individuals affected in the prime of their life) is different from high-income countries. As such, HF is now responsible for 7-10% of medical admissions in the region. (7) These are entirely based on studies on acute HF. There are only few data on chronic HF in Africa. Furthermore, the nexus between endemic infections such as tuberculosis (TB) and HIV/AIDS and other non-communicable or non-infectious risk factors and HF in Africa is scarcely documented.

Gaps in knowledge on heart failure in sub-Saharan Africa

1. Co-morbidities in HF patients, which are common and important to outcomes, have not been well studied in large cohorts in sub-Saharan Africa (SSA).
2. The role and co-occurrence of infection such as tuberculosis and HIV /AIDS has not been extensively explored in the region.

4 There is paucity of information on the long-term outcome of HF in SSA (rehospitalization and mortality) 5 Current phenotypes of HF (HFrEF, HFpEF, HFmrEF), their clinical and sociodemographic predictors, management and outcomes are not well described in SSA.

6 There is also paucity of data on the assessment of barriers to HF care in SSA.

7 Significantly, given its potential enormous cost implications (both related to direct health care costs and economic burden on affected individuals and their families) there is virtually no data on the economic burden of HF in SSA.

8 There is paucity of data on cultural and social conceptions of heart failure in SSA.

9 There are few genetic and genomic HF studies in sub-Saharan Africa especially in Nigeria (the region's most populous country).

10 We do not know to what extent are standard care pathways and evidence-based treatment algorithms applied in the management of HF Ibadan. We also do not know to what extent high out of pocket expenses contribute to low levels of treatment. Furthermore, we do not know the scope for quality improvement to improve outcomes and reduce mortality rates in Nigeria.

11 Although there is existing evidence of economic cost and impact from the Abeokuta HF registry, data on catastrophic healthcare spending linked to CHF care from a household perspective are lacking. In addition, the extent to which out of pocket costs (drugs and consultations/ admissions) act as a barrier to continuing evidence-based care is not available.

12 Lastly the extent patient-centred approaches (their values and preference) are applied to care plans in Ibadan is not available. The use of patient-reported outcome measures in routine care (PROMs) has not been explored.

Aim The primary objective of this study is to assess the long-term outcomes, risk factors, clinical phenotypes, and genomics of HF in Ibadan, Nigeria, estimate catastrophic healthcare cost associated with CHF and how it affects evidence-based care; understand cultural and social conceptions of HF in the city and by extension in Nigeria Objectives

1. To define the clinical profile of heart failure in Ibadan, Nigeria
2. To determine the short-term, medium-term and long-term outcome of heart failure in Ibadan and by extension in Nigeria.
3. To identify comorbidities (Infections and non-infections) in heart failure in Nigeria and the clinical implications
4. To develop predictive models of mortality, rehospitalization and complications associated with heart failure in Nigeria.
5. To estimate the catastrophic healthcare cost of HF in Ibadan
6. To develop a community engagement and education programmes on non-communicable diseases (NCDs).
7. To explore the cultural and social conceptions of heart failure in Ibadan, Nigeria.
8. To investigate genetic associations of ACE, LMNA and Troponin T (TNNT2) variants with HF in the study population METHODS Study design The study shall be prospective study. It is expected that about 2500-3000 subjects with HF shall be recruited over a 5-year period and followed up at 6, 12, 24 months and five years.

Study location The study shall be conducted at the University College Hospital, Ibadan, Nigeria. The University College Hospital, Ibadan is the oldest teaching hospital in Nigeria and affiliated to the University of Ibadan. Currently the hospital has over 950 bed spaces and 163 examination couches and a current bed occupancy rate of 55-60%. The hospital has over 60-clinical departments. It serves a population of over 10million people and receives referrals from all over the country and as well from the West African sub-region.

Inclusion and exclusion criteria Subjects are eligible to participate if they are 18 years and older and have clinically and echocardiographically confirmed HF.

Data collection and case definition Data from each subject shall be obtained using a uniform and standardized case report forms (CRF). A detailed clinical documentation on cases of HF will be undertaken. The following data shall be obtained: study identification number, demographic data, date of diagnosis of HF and pre-admission history (previous heart failure related admissions). Others include NYHA functional class, symptoms, signs, self-reported cardiovascular risk factors, aetiology of HF, co-morbidities, blood investigations, point of care biomarker, Chest X-ray, 12-lead ECG, echocardiography, medications, barriers to care, quality of life data etc.

Case definition The European Society of Cardiology guideline shall be employed for the diagnosis of HF. All cases shall be confirmed at echocardiography. All the echocardiograms shall be performed by trained personnel. The quality assurance information of the procedure at Ibadan has been published.

Blood Collection and Testing Blood sample will be obtained during the enrolment visit and shipped to the central laboratory at Ibadan for analysis of biochemical biomarkers, including risk factors for HF and related cardiovascular diseases.

Follow-up Follow-up of subjects shall be through clinic visits or via telephone. Telephone numbers of next of kin of patients shall also be obtained. Information that shall be obtained during the follow-up period shall include amongst others: well-being of the patient, symptoms, signs, medications as well as well as events such as readmission, deaths etc.

Deaths shall be recorded and their cause shall be ascertained by the review of various source documents or verbal autopsy to classify the cause of death.

Medication Adherence Questions regarding medication adherence will be asked at baseline and 1-year visit. This medication adherence questionnaire will ask questions on how often patients take their HF medicines, what factors/events may lead to their missing medicines, and reasons why they may miss medications.

Capture of dietary Questionnaire Dietary questionnaire shall be administered on the patients. This will be used to collect information about the type, portion size, quantity and frequency of commonly consumed foods. This will incorporate validated nutritional information in Nigeria.

Economic cost analysis Healthcare costs shall be estimate for one year in the Nigerian Naira and will be converted to US Dollar [$US] at the prevailing exchange rate at the time of the study. Catastrophic healthcare spending (CHS) occurs when out-of-pocket payments is above a given percentage of households' total income/total expenditure. Three thresholds, 10%, 20% and 40% will be applied to ascertain the burden of catastrophic healthcare spending among patients' household level.

Sample size calculation Though this study is prospective in design, it is largely exploratory because most of the objectives are descriptive in nature. For a descriptive study, a sample size of 400 is sufficient to estimate the level of any outcome with 95% confidence. However, to make adequate allowance for study objectives that requires comparisons, we plan to recruit at least of 1500-2000 patients.

Statistical analysis All variables will be summarised using appropriate descriptive statistics. Means and proportions will be estimated with two-tailed 95% confidence intervals. Specified patients' outcomes will also be summarised using proportions. Factors associated with patients' outcomes will be investigated using multivariable logistic regression models. Crude and adjusted Odds Ratio (OR) with 95% confidence intervals (CI) will be estimated Ethical considerations Ethical standard The Ibadan Acute and Chronic Heart Failure Project will be conducted in full compliance with the principles of the Declaration of Helsinki or with the laws and regulations of Nigeria.

Data management and statistical analysis Categorical variables shall be displayed as frequencies and proportions. Group comparison shall be done with the student's t-test and Chi square statistics shall be used for comparison of categorical variables. Survival function estimates shall be performed using the Kaplan-Meier method and the difference shall be tested using log-rank test. The follow up shall be censored at 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

All cases of heart failure

Exclusion Criteria:

No consent to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults aged 18-100 years presenting with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5 years
  All cause mortality

SECONDARY OUTCOMES:
Hospitalisation | 5 years
  Hospital readmission

CONTACTS AND LOCATIONS:
Overall Officials: Okechukwu S Ogah, PhD, Principal Investigator — Cardiology Unit, Department of Medicine, University College Hospital Ibadan, Nigeria
Locations (1):
- University College Hospital Ibadan, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No
There is no plan for this

REFERENCES:
- [Result] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Result] Cowie MR, Mosterd A, Wood DA, Deckers JW, Poole-Wilson PA, Sutton GC, Grobbee DE. The epidemiology of heart failure. Eur Heart J. 1997 Feb;18(2):208-25. doi: 10.1093/oxfordjournals.eurheartj.a015223. No abstract available. PMID 9043837
- [Result] Bui AL, Horwich TB, Fonarow GC. Epidemiology and risk profile of heart failure. Nat Rev Cardiol. 2011 Jan;8(1):30-41. doi: 10.1038/nrcardio.2010.165. Epub 2010 Nov 9. PMID 21060326
- [Result] Redfield MM, Jacobsen SJ, Burnett JC Jr, Mahoney DW, Bailey KR, Rodeheffer RJ. Burden of systolic and diastolic ventricular dysfunction in the community: appreciating the scope of the heart failure epidemic. JAMA. 2003 Jan 8;289(2):194-202. doi: 10.1001/jama.289.2.194. PMID 12517230
- [Result] Mosterd A, Hoes AW, de Bruyne MC, Deckers JW, Linker DT, Hofman A, Grobbee DE. Prevalence of heart failure and left ventricular dysfunction in the general population; The Rotterdam Study. Eur Heart J. 1999 Mar;20(6):447-55. PMID 10213348
- [Result] Damasceno A, Mayosi BM, Sani M, Ogah OS, Mondo C, Ojji D, Dzudie A, Kouam CK, Suliman A, Schrueder N, Yonga G, Ba SA, Maru F, Alemayehu B, Edwards C, Davison BA, Cotter G, Sliwa K. The causes, treatment, and outcome of acute heart failure in 1006 Africans from 9 countries. Arch Intern Med. 2012 Oct 8;172(18):1386-94. doi: 10.1001/archinternmed.2012.3310. PMID 22945249
- [Result] Ogah OS, Stewart S, Falase AO, Akinyemi JO, Adegbite GD, Alabi AA, Ajani AA, Adesina JO, Durodola A, Sliwa K. Contemporary profile of acute heart failure in Southern Nigeria: data from the Abeokuta Heart Failure Clinical Registry. JACC Heart Fail. 2014 Jun;2(3):250-9. doi: 10.1016/j.jchf.2013.12.005. Epub 2014 Apr 30. PMID 24952692